CLINICAL TRIAL: NCT03010046
Title: A Phase 1, Randomized, Placebo-controlled, Double Blind, Single, Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ANX005 Monotherapy and ANX005 in Combination With IVIg in Healthy Volunteers
Brief Title: Single Dose Study of ANX005 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: ANX005 well tolerated at doses studied; study discontinued and initiated in patient population
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANX005-CP01
Record Dates: First submitted 2016-12-21; First posted 2017-01-04 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Safety and Tolerability in Healthy Volunteers
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ANX005 Monotherapy (Experimental): ANX005 intravenous infusion
  Interventions: Drug: ANX005
- ANX005 and IVIg Combination Therapy (Experimental): ANX005 intravenous infusion in combination with intravenous immunoglobulin (IVIg)
  Interventions: Drug: ANX005; Drug: IVIg
- Placebo (Placebo Comparator): Placebo intravenous infusion
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: ANX005 — Single ascending dose intravenous infusion
  Arms: ANX005 Monotherapy; ANX005 and IVIg Combination Therapy
Drug: IVIg — IVIg infusion in Cohorts 4b and 5b only. Randomized to ANX005 followed by IVIg or placebo followed by IVIg.
  Arms: ANX005 and IVIg Combination Therapy
Drug: Placebos — 0.9% saline intravenous infusion
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, ascending, single-infusion, sequential group study. Single, ascending doses will be administered to approximately 64 subjects, with an option for 1 additional multi-dose cohort in approximately 8 subjects. The primary objective is to evaluate the safety of ANX005 administered as an intravenous infusion as a single agent and in combination with intravenous immunoglobulin (IVIg). The optional multi-dose cohort will evaluate either additional subjects at the maximum tolerated dose or ANX005 administered as 2 infusions.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 years and older
* Females must be postmenopausal, surgically sterilized, or willing and able to use 2 methods of contraception throughout the study and for 1 month after the final study visit
* Willing and able to undergo vaccination if not vaccinated recently

Exclusion Criteria:

* History of any autoimmune disease, meningitis, septicemia or pneumonia
* History of hypercoagulable diseases, hyperviscosity, thrombosis, renal dysfunction or acute renal failure
* Known genetic deficiencies of the complement cascade system
* History of conditions whose symptoms and effects could alter protein catabolism or IgG utilization, e.g. protein-losing enteropathies or nephrotic syndrome
* Body weight less than 50 kg or greater than 100 kg
* Hypersensitivity or allergic reactions to any excipients in the ANX005 drug product
* (Cohorts 4b and 5b) Known selective IgA deficiency or presence of antibodies to IgA at screening
* (Cohorts 4b and 5b) Prior reaction or hypersensitivity to blood products, including IVIg or any of the excipients in IVIg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events as assessed by CTCAE v4.03 | Day 43
  Safety is assessed throughout the study. Day 43 is the last visit.

SECONDARY OUTCOMES:
Peak plasma concentration | Day 43
Determine effective dose of ANX005 | Day 43
  Percent of subjects with a biologic response, defined as a reduction of serum CH50 percent change from baseline at 21 and 28 days after the first ANX005 infusion
Area under the plasma concentration versus time curve (AUC) | Day 43
Terminal half-life | Day 43

OTHER OUTCOMES:
Explore relationship of AUC with PD responses in serum | Day 43
Explore relationship of AUC with PD responses in CSF | Day 43
Explore relationship of half-life with PD responses in serum | Day 43
Explore relationship of half-life with PD responses in CSF | Day 43

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Calman, MD, Study Director — Annexon Medical Monitor; Jason Lickliter, MBBS PhD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lansita JA, Mease KM, Qiu H, Yednock T, Sankaranarayanan S, Kramer S. Nonclinical Development of ANX005: A Humanized Anti-C1q Antibody for Treatment of Autoimmune and Neurodegenerative Diseases. Int J Toxicol. 2017 Nov/Dec;36(6):449-462. doi: 10.1177/1091581817740873. Epub 2017 Dec 4. PMID 29202623